CLINICAL TRIAL: NCT05462145
Title: A Prospective, Multicenter Clinical Study to Evaluate the Safety and Effectiveness of the Globe® Pulsed Field System for Treating Patients With Symptomatic Paroxysmal or Persistent Atrial Fibrillation
Brief Title: Safety and Effectiveness of the Globe® Pulsed Field System for Treating Patients With Symptomatic Paroxysmal or Persistent Atrial Fibrillation
Acronym: PULSAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kardium Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOC-189367
Record Dates: First submitted 2022-07-13; First posted 2022-07-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
Keywords: Pulsed Field Ablation; Irreversible Electroporation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Globe Pulsed Field System (Experimental)
  Interventions: Device: Globe Pulsed Field System

INTERVENTIONS:
Device: Globe Pulsed Field System — Ablation and atrial mapping with the Globe Pulsed Field System

SUMMARY:
This study will evaluate the safety and effectiveness of the Globe® Pulsed Field System for treating patients with symptomatic paroxysmal or persistent atrial fibrillation (AF).

ELIGIBILITY:
Key inclusion criteria:

* A diagnosis of recurrent symptomatic paroxysmal or persistent AF
* Failure or intolerance of at least one antiarrhythmic drug (AAD) Class I or III

Key exclusion criteria:

* Long-standing persistent AF (sustained >12 months)
* Atrial fibrillation secondary to a reversible cause or of non-cardiac origin
* History of thromboembolic events within the past six months
* Myocardial infarction (MI)/percutaneous coronary intervention (PCI) within the last three months
* Any cardiac surgery within the previous six months
* Prior left atrial ablation or surgical procedure
* Presence of an implanted cardiac device
* Body mass index (BMI) >40 kg/m^2
* Left ventricular ejection fraction (LVEF) <35%
* Anterior-posterior left atrial (LA) diameter >55mm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Effectiveness endpoint | 12 months
  Number of subjects with freedom from documented atrial fibrillation, atrial flutter, and atrial tachycardia (AF/AFL/AT) 12 months post-procedure.
Safety endpoint | 7 days
  Rate of subjects presenting with one or more of the specified primary safety events within 7 days of the index ablation procedure.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (12):
  - Grandview Medical Center, Birmingham, Alabama
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - Sutter Health - California Pacific Medical Center, San Francisco, California
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Mercy Hospital, Miami, Florida
  - Johns Hopkins, Baltimore, Maryland
  - Beaumont Hospital, Royal Oak, Michigan
  - Mt. Sinai Hospital, Guggenheim Pavilion, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
- Canada (2):
  - St.Paul's Hospital, Vancouver, British Columbia
  - McGill University Health Centre, Montreal, Quebec
- Motol and Homolka University Hospital, Prague, Czechia
- Germany (3):
  - Heart and Diabetes Center NRW, Bad Oeynhausen
  - Charité Campus Virchow Clinic, Berlin
  - Westpfalz-Klinikum GmbH Kaiserslautern, Kaiserslautern

REFERENCES:
- [Background] Reddy VY, Kottkamp H, Calkins H, Nair DG, Sommer P, Hussein AA, Schumacher B, Dukkipati S, Neuzil P, Oza S, Woods C, Deyell MW, Osorio J, Verma A; PULSAR Investigators. Pulsed-Field Ablation to Enhance the Durability of Pulmonary Vein Isolation and Treat Paroxysmal Atrial Fibrillation. J Am Coll Cardiol. 2026 Jan 14:S0735-1097(25)10256-8. doi: 10.1016/j.jacc.2025.10.084. Online ahead of print. PMID 41563170